CLINICAL TRIAL: NCT03828240
Title: HIP Fracture REhabilitation Programme for Elderly With Hip Fractures
Acronym: HIP-REP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Municipality of Herlev (Unknown); Municipality of Lyngby-Taarbæk (Unknown); Municipality of Gentofte (Unknown); Copenhagen University Hospital at Herlev (Other); Jonkoping University (Other); Intersectoral Research Unit (Unknown); Metropolitan University College (Other); Danish Association of Occupational Therapist (Other); Danish Regions Development and Research (Unknown)
Responsible Party: Principal Investigator, Carsten Bogh Juhl, Principal Investigator, Herlev and Gentofte Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HerlevGentofte
Record Dates: First submitted 2019-01-29; First posted 2019-02-04 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: Activity-based intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enhanced rehabilitation (Other)
  Interventions: Other: HIP fracture REhabilitation Programme for the elderly with hip fractures

INTERVENTIONS:
Other: HIP fracture REhabilitation Programme for the elderly with hip fractures — Eight-week activity-based intervention for elderly with hip fractures; one intervention during the hospital stay, four interventions at the elderly's municipality.

SUMMARY:
Objectives: To evaluate the feasibility of a HIP fracture REhabilitation Programme (HIP-REP).This study will investigate adherence, satisfaction, technical and practical circumstances regarding implementation and taking this into account when evaluating the feasibility of the HIP-REP program.

Hypothesis: By testing the feasibility of a HIP-REP for the participants and the usefulness of the selected measurement tools, the investigators will be able to evaluate and adjust the HIP-REP before evaluating this in a larger Randomized controlled trial (RCT).

DETAILED DESCRIPTION:
Little is known about the feasibility and effect of an intersectoral rehabilitation intervention aiming at reducing the decrease in Activities of Daily Living (ADL) ability for elderly with hip fractures. Despite positive surgical outcomes, one-quarter dies within a year after surgery, around eight percent are readmitted to hospital, and just one-third regain their pre-fracture level of physical functioning and ADL ability. After hip fracture, the loss of independence, and further decrease in ADL ability often persists beyond three months after surgery. This increases the risk of social isolation, depression and thus a decrease in Quality of Life (QoL). Therefore, the investigators want to evaluate whether an activity-based rehabilitation intervention across sectors is feasible and influences this fragile group of patients. The investigators hope to increase the ability to safely and independently perform ADL in elderly with hip fractures, and thereby enhance their health-related QoL.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Recent proximal hip fracture (S 72.0 Medial femur fracture, S 72.1, Pertrochanteric femur fracture, S 72.2 Subtrochanteric femur fracture)
* Living at home prior to hip fracture in Herlev, Gentofte or Lyngby-Taarbæk municipalities
* Ability to give informed consent
* Discharged from hospital and receiving or having received rehabilitation in one municipalities within the last 3 months from onset

Exclusion Criteria:

* Not expected to be discharged to home or rehabilitation centers in the municipality
* Not able to speak and/or understand Danish
* Have prior severe physical and /or mental disabilities

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Motor and Process Skills | Change from baseline at motor and process skills 3 months after baseline testing
  The assessment measures the quality of a person's activity of daily living task performance. An observational assessment that allows for evaluation of change in motor and process skills and their effect on the ability of an individual to perform complex or instrumental and personal activities of daily living. The instrument consists of 16 motor and 20 process skill abilities that are rated on a 4-point scale, In all, 36 discrete ratings of motor and process skills are made during observation.

SECONDARY OUTCOMES:
European Quality of Life Questionnaire | at baseline and 3 months after baseline testing
  A survey collecting information about health related quality of life comprising five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Verbal Rating Scale | at baseline and 3 months after baseline testing
  An assessment measuring the intensity of pain. The patient chooses one of those: none, mild, moderate or severe.
Occupational Balance Questionnaire | at baseline and 3 months after baseline testing
  An assessment that measures the patients satisfaction with the amount and variation of occupations; . It consists of 13 items measured on six-step ordinal scales. The patient chooses one of those: Disagree, partly disagree, partly agree or agree.
Satisfaction with daily occupations | at baseline and 3 months after baseline testing
  An instrument measuring satisfaction with everyday occupations addressing four areas of everyday occupations: work and work-related occupations, leisure occupations, domestic occupations and self-care. The patient chooses on a scale from 1 to 7. 1 = Not satisfied to 7 = Very satisfied.
Cumulated Ambulation Score | at baseline
  The Cumulated Ambulation Score is evaluating patients' basic mobility (getting in and out of bed, sit-to-stand from a chair and walking). Each of the three activities is scored from 0-2, resulting in a daily score of 0-6.
New Mobility Score | at baseline and 3 months after baseline testing
  The New Mobility Score is a composite score of the patient's ability to perform: indoor walking, outdoor walking and shopping, providing a score between zero and three (0: not at all, 1: with help from another person, 2: with an aid, 3: no difficulty) for each function, resulting in a total score from 0 to 9, with nine indicating a high prefracture functional level.
Functional Recovery Score | at baseline and 3 months after baseline testing
  Functional Recovery Score assess the level of function with eleven-items comprised of three main components: basic activities of daily living assessed by four items, instrumental activities of daily living assessed by six items, and mobility assessed by one item. Basic activities of daily living comprise 44 percent of the score; instrumental activities of daily living comprise 23 percent, and mobility comprises 33 percent. Complete independence in basic and instrumental activities of daily living and mobility results in a score of 100 percent.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy and Occupational Therapy, Copenhagen University Hospital, Herlev and Gentofte, Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ropke A, Morville AL, Moller TE, Delkus ECG, Juhl CB. HIP Fracture REhabilitation Program for older adults with hip fracture (HIP-REP) based on activity of daily living: a feasibility study. BMC Geriatr. 2022 Apr 27;22(1):370. doi: 10.1186/s12877-022-03039-x. PMID 35477380
- [Derived] Ropke A, Lund K, Thrane C, Juhl C, Morville AL. Developing an individualised cross-sectoral programme based on activities of daily living to support rehabilitation of older adults with hip fracture: a qualitative study. BMJ Open. 2021 Jun 18;11(6):e044539. doi: 10.1136/bmjopen-2020-044539. PMID 34145009